CLINICAL TRIAL: NCT03443999
Title: Prospective Evaluation of the Supraflex Family Sirolimus-eluting Coronary Stent System in a 'Real-World' Patient Population
Brief Title: S-FLEX Netherlands Registry: Prospective Evaluation of the Supraflex Family Sirolimus-eluting Coronary Stent System
Status: Recruiting | Type: Observational
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: SFLX/Netherlands/001
Record Dates: First submitted 2018-02-16; First posted 2018-02-23 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Sirolimus-eluting Stent; Biodegradable Polymers
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Supraflex Family Sirolimus-eluting Coronary Stent System — Patient implanted with at least one Supraflex Family sirolimus-eluting stent as a part of planned clinical care

SUMMARY:
The primary objective of this registry is to evaluate the safety and efficacy of the Supraflex Family sirolimus-eluting coronary stent system in a 'real-world' patient population requiring stent implantation.

DETAILED DESCRIPTION:
To overcome the potential drawback of the durable polymer a new generation of drug-eluting stent (DES) with a biodegradable polymer has been designed. The first-generation sirolimus-eluting or paclitaxel-eluting stents have a polymer release of antiproliferative drugs from a stainless steel stent platform. More recently, second generation DES have been developed not only to improve long-term DES safety but also to facilitate the procedure by using a cobalt-chromium (Co-Cr) stent platform. Co-Cr is stronger and more radiopaque than stainless steel, and thus allows strut thickness and total stent volume to be reduced while maintaining radial strength leading to a more flexible and deliverable stent platform.

The Sahajanand Medical Technologies Pvt. Ltd. (SMT) has developed sirolimus-eluting stent that contain a biodegradable polymer coating and a Co-Cr stent platform. The purpose of this registry is to evaluate the Supraflex Family sirolimus-eluting stent in a 'real-world' patient population, in order to determine the safety and efficacy of the stent in wider usage.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. The patient, or legal representative, has been informed of the nature of the registry and has consented to participate and authorised the collection and release of his/her medical information by signing a Patient Informed Consent Form
3. Treating physician has electively implanted at least one Supraflex Family stent as part of the patient's planned clinical care.
4. The patient is willing and able to cooperate with study procedures and required follow up visits

Exclusion Criteria:

1. Women with known pregnancy or who are lactating
2. High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
3. Currently participating in another study that has not completed the primary endpoint or that clinically interferes with the current registry requirements
4. Planned surgery within 6-month of PCI unless dual anti-platelet therapy is maintained throughout the peri-surgical period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-world patient population assigned for PCI who present with at least one angiographically documented coronary artery lesion suitable for percutaneous treatment with implantation of Supraflex Family sirolimus-eluting stent.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  TLF defined as a composite of cardiac death, target vessel myocardial infarction (Q wave and non-Q wave), or clinically-driven target lesion revascularization (TLR) by percutaneous or surgical methods.

SECONDARY OUTCOMES:
Target Vessel Failure (TVF) | 12 months
  TVF defined as a composite endpoint of cardiac death, target vessel myocardial infarction, or clinically-driven target vessel revascularization (TVR)
Major Adverse Cardiac Events (MACE) | 12 months
  MACE defined as a composite endpoint of cardiac death, myocardial infarction (Q wave and non-Q wave), emergent coronary bypass surgery, or repeat target lesion revascularization (clinically driven/clinically indicated) by percutaneous or surgical methods
Stent Thrombosis | 12 months
  Stent thrombosis rates according to ARC classification
All Deaths | 12 months
  Cardiac death and non-cardiac death (vascular and non-cardiovascular)
Any Myocardial Infarction (MI) | 12 months
  Q wave and non-Q wave MI
Any Repeat Revascularization | 12 months
  Target lesion revascularization (TLR) and target vessel revascularization (TVR)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. A.J.J. IJsselmuiden, MD., Principal Investigator — Amphia Hospital, Breda, The Netherlands
Locations (7):
- Netherlands (7):
  - Amphia Ziekenhuis, Breda, North Brabant
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Tergooi Ziekenhuis, Blaricum, North Holland
  - Medical Center Leeuwarden, Leeuwarden, Provincie Friesland
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - ZorgSaam Hospital, Terneuzen, Zeeuws- Vlaanderen

IPD SHARING:
Plan to Share IPD: No